CLINICAL TRIAL: NCT03105388
Title: STOP-BANG Score and Cephalometry in Prediction of Difficult Airway in Patients at Risk of Obstructive Sleep Apnoea
Brief Title: STOP-BANG and Cephalometry in Prediction of Difficult Airway in Patients at Risk of OSA
Status: Completed | Type: Observational
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Rhendra Hardy Mohamad Zaini, Senior consultant anesthetist and lecturer, Universiti Sains Malaysia
Other Study IDs: USM/JEPeM/15010010
Record Dates: First submitted 2017-03-09; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Sleep Apnea; Difficult Intubation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Incidence of difficult laryngoscopy and difficult intubation are higher among patients with obstructive sleep apnoea (OSA). Precision in making the diagnosis and predicting difficult laryngoscopy preoperatively may help to reduce anesthetic complications. This study was designed to evaluate the diagnostic performance of combined and non-combined radiological parameter (mandibulohyoid distance) and STOP-BANG questionnaire as screening tool.

.

Methodology:

Forty-one subjects who were at risk of OSA, undergoing general anaesthesia will be included using STOP-BANG questionnaire. Mandibulohyoid distance and other radiological parameters will be measured from lateral cephalometry. Evaluation for difficult laryngoscopy will be carried out during anaesthesia.

DETAILED DESCRIPTION:
RESEARCH DESIGN:Cross sectional study

STUDY HYPOTHESES: There is a significant correlation between STOP-BANG score and cephalometric measurement with difficult intubation in patients at risk of Obstructive Sleep Apnoea.

Null hypothesis:

There is no significant correlation between STOP-BANG score and cephalometric measurement with difficult intubation in patients at risk of Obstructive Sleep Apnoea.

SAMPLE SIZE ESTIMATION This is a cross sectional study with 2 means. For objective 1, sample size calculation is done using power and sample size program version 3.1.2

* Population Standard deviation for STOP-BANG score according to Graciela E.Silva et al. ,2011 is 1.3, and the estimated difference from population mean is 1.28 with 95% confidence, Z is 1.96 , power of study 0.8
* Estimated Sample size required is 34.
* With 20% drop out rate , 34+(34x0.2)=41
* Sample size required is 41

For objective 2, sample size calculation using PS program version 3.1.2, Population Standard deviation for mandibular-hyoid distance is 0.7 according to A.S.Hiremath et al., 1998 and the estimated difference from population mean is 0.68 with 95% confidence, Z is 1.96 . power of study 0.8

* Estimated Sample size required is 34.
* With 20% drop out rate , 34+(34x0.2)=41
* Sample size required is 41

For objective 3, sample size calculation was done using G power 3.1.9.2 program.

* Based on expert opinion, the expected correlation between STOP-BANG score and cephalometric measurement (mandibulohyoid distance) is at least 0.60 confidence interval of 95%. Power of study 0.8.
* The required sample size is 30.
* Expected 10% of dropout rate.
* 30+(30x 0.1)= 33

For objective 4, sample size calculation using PS size program version 3.1.2,

* Population SD for age is 12.3 according to Sang Jun Lee et al., 2011, and the estimated difference from population mean is 12.25 with 95% confidence, Z is 1.96 . power of study 0.8
* Estimated Sample size required is 34.
* With 20% drop out rate , 34+(34x0.2)=41
* Sample size required is 41
* Population SD for height is 6.9 according to Sang Jun Lee et al., and the estimated difference from population mean is 6.85 with 95% confidence, Z is 1.96 .power of study 0.8
* Estimated Sample size required is 34.
* With 20% drop out rate,
* Sample size required is 41
* Population SD for weight is 9.7 according to Sang Jun Lee et al, and the estimated difference from population mean is 9.65 with 95% confidence, Z is 1.96. Power of study 0.8
* Estimated Sample size required is 34.
* With 20% drop out rate,
* Sample size required is 41
* Population SD for BMI is 3.2 according to Sang Jun Lee et al., and the estimated difference from population mean is 3.15 with 95% confidence, Z is 1.96 .power of study 0.8
* Estimated Sample size required is 34.
* With 20% drop out rate,
* Sample size required is 41
* Population Standard deviation for neck circumference is 3.7 according to Sang Jun Lee et al, and the estimated difference from population mean is 3.65 with 95% confidence, Z is 1.96. power of study 0.8
* Estimated Sample size required is 34.
* With 20% drop out rate,
* Sample size required is 41

Thus the highest number of sample size 41 is taken.

SAMPLING METHODS All patients at risk of OSA who come for elective surgery and fulfilled the selection criteria are included.

RECRUITMENT OF SUBJECT AND INFORMED CONSENT SEEKING All patients who come for elective surgery under general anesthesia and at risk of Obstructive Sleep Apnea will be screened using STOP-BANG questionnaires .Those that fulfilling the selection criteria will be recruited.

Written informed consents were obtained one day before the operation day. Sleep study not part of the objective of this study. Consent will be taken one day before the operation day. Patients will receive explanation about the objectives of the study, one lateral head and neck x-ray will be taken one day before operation, while other procedures will match the standard procedure. Normal laryngoscopy will be done to assess their airway using the Cormack Lehance scoring, then they will be intubated using videolaryngoscope.

STUDY AREA Operation theater of Hospital Universiti Sains Malaysia.

CONFLICT OF INTEREST This study is done for the benefit of patient. There is no conflict of interest.

All patients who come for elective surgery under general anesthesia and at risk of Obstructive Sleep Apnea will be screened using STOP-BANG questionnaires .Those who are fulfilling the selection criteria will be recruited.

Written informed consents were obtained one day before the operation day.

PRIVACY AND CONFIDENTIALITY

* Patient's medical information will be kept confidential by the study doctor and staff and will not be made publicly available unless disclosure is required by law.
* Data obtained from this study that does not identify patient individually will be published for knowledge purposes. Patient's original medical records may be reviewed by the researcher, the Ethical Review Board for this study and regulatory authorities for the purpose of verifying clinical trial procedures and/or data. Patient's medical information may be held and processed on a computer.

PROPOSED DATA ANALYSIS Group A for whom the intubation is easy, is limited to the patients with a Cormack Lehance grade of 1 and 2 ( the glottis is immediately visible).

Group B for whom the intubation is difficult would comprise of patients given a Cormack Lehance grade of 3 and grade 4( poor visibility of the glottis).

All of the values are shown as mean +/- SDs and as percentages. Independent sample t-test , cross-tabulation and chi square test are used for comparing the two groups.

P values <0.05 are considered significant. A comprehensive evaluation is done by binary logistic regression analysis and a multivariate test to see the effects of each independent variable on the dependent variables.

STUDY PROTOCOL Human ethical approval was obtained from HUSM's ethics committee to do the study.

41 ASA class I and II (normal healthy patient or mild systemic disease) requiring general anesthesia, with age range between 18 year old to 75 year old will be recruited. Preoperatively, each patient will be interviewed by a research resident who completed the first study questionnaire regarding the diagnosis of OSA, based on self- report by the patient. For patients not previously tested/ diagnosed for OSA, the STOP-BANG questionnaire will be used to determine a STOP-BANG score.

In the STOP questionnaire 4 will be used to construct the STOP score:

* Snore is considered affirmative if the participant reported snoring loudly (louder than talking or loud enough to be heard through closed doors).
* Tiredness/sleepy during the day is affirmative if the participant reported yes to feeling unrested during the day no matter how many hours of sleep he/she had (often and almost always = yes; never, rarely, and sometimes = no) and reported feeling tired (all of the time, most of the time, a good bit of the time = yes, and some of the time, a little bit of the time, and none of the time = no).
* Observed stop breathing is defined as yes if participant answered affirmative to the question "based on what the participant have noticed or household members have told them, are there times when they stop breathing during their sleep?"
* Blood Pressure is defined as positive if the participant answered yes to being treated with medication for high blood pressure.

The BANG portion will be evaluated by assessing:

* Body mass index (BMI > 35 kg/m2)
* Age (over 50 years old)
* Neck circumference (neck circumference > 40 cm)
* Gender (male).

One point was assigned for each affirmative answer; 0 for no answers.

A STOP-BANG score of ≥ 3 affirmative is chosen for this study, as this score had a very high sensitivity and negative predictive value for moderate/severe OSA, and had been suggested as a good cutoff value for high OSA prevalence among surgical populations such as bariatric patients (Chung et al 2012.)

The investigators exclude pregnant patients, those who were not fasted for at least 6 hours prior to anesthesia, and those with GERD.

The patient's age, gender, ASA status, height, weight, BMI, Thyromental distance, and neck circumference are recorded.

The patient will be made to sit up and stick out their tongue as far as they could, in order to observe the internal structure of the pharynx under lighting. The findings can be classified using the Mallampati scoring systems.

Mallampati et al. classified the pharyngeal structure into 3 types, but Samsoon and Young created a Modified Mallampati Test that divides the structure into 4 types .

* Class 1 is when the soft palate, the fauces, the uvula and the anterior and posterior tonsillar pillars are visible.
* Class II is where all the class I structures are visible except for the tonsillar pillars.
* Class III is where only the base of the uvula is visible.
* Class IV is where the uvula cannot be seen and only the soft palate is visible.

After clinical assessment, Lateral Cephalometry (lateral head and neck x-ray) will be taken in a neutral head position in radiological department. Mandibular-hyoid distance will be measured.

Patients will be well fasted overnight before the operation. No premedication with sedative effects will be given on the operation day.

Standard monitoring include: ECG, non-invasive automatic blood pressure monitoring, pulse oximeter. The blood pressure and pulse rate will be taken before induction of anesthesia.

Anesthesia will be performed by a skilled anesthesiologist who is not the investigator for this study, and do not know the cephalometric measurement of the patient.

Pre-oxygenation will be using 100% oxygen 5 L/ min for 2-3 min given a by a mask and this was inspired by voluntary respiration.

IV Fentanyl 1.5-2mcg per kg and IV Propofol 1-2mg per kg, will be administrated in titration. After loss of consciousness, 0.9 mg/kg IV Rocuronium ( a muscle relaxant) will be given. When the state of muscle relaxation is observed, guided by TOF nerve stimulator, the head will be placed in the sniffing position to facilitate intubation. Then a size 3 curved laryngoscopy will be use to maximize exposure of the glottis, and without pressing the thyroid cartilage, the airway will be evaluated and graded following Cormack and Lehance grading system.

Cormack Lehane proposed grading the laryngoscopic view from grade I to grade.

* Grade I is when the epiglottis and vocal cords are completely exposed.
* Grade II is when only rear of the vocal cords can be seen.
* Grade III is when only the epiglottis is exposed.
* Grade IV is when only the soft palate can be seen.

Subsequently patient will be intubated using videolaryngoscope and with appropriate ETT size. In standard practice , all patients will be intubated using conventional laryngoscopy, but in our study , they will be intubated using videolaryngoscope which is a device to assist in difficult intubation.

After intubation, mechanical ventilation will be performed with oxygen at 2L/min , with the tidal volume 8ml/kg and the tidal rate 12 bpm. Anesthesia will be maintained with inhalational agent Sevoflurane at the MAC of 1.

After surgery, all patients will be reversed using Suggammadex (a specific antidote for Rocuronium) or standard reversal drugs mixture (1 mg atropine and 2.5 mg neogstigmine), this was according to standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patient of age 18 years old and above.
* American Society of Anesthesiologist (ASA) physical status I and II.
* Age range (18- 75yo).
* Operation requiring general anesthesia
* All patient at risk of Obstructive Sleep Apnea with STOP-BANG questionnaire scoring ≥ 3 positive response are selected on the day of admission.

Exclusion Criteria:

* Pregnant patient.
* Not fasted as least for 6 hours
* Has gastroesophageal reflux.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who come for elective surgery under general anesthesia and at risk of Obstructive Sleep Apnea will be screened using STOP-BANG questionnaires.Those who are fulfilling the selection criteria will be recruited.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Correlation between STOP-BANG score and Cormack Lehance view. | May 2015 - February 2016
  STOP-BANG score (Snoring, Tired during daytime, Observed apnoea, High blood pressure, BMI, Age, Neck circumference: Neck circumference, Gender)

SECONDARY OUTCOMES:
Correlation between Mandibular-hyoid distance and Cormack Lehance view. | May 2015 - February 2016
  Correlation between Mandibular-hyoid distance (mm), measure from lateral cephalometry and Cormack Lehance view.

CONTACTS AND LOCATIONS:
Overall Officials: Rhendra Hardy Mohd Zaini, MD, MMed, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hiremath AS, Hillman DR, James AL, Noffsinger WJ, Platt PR, Singer SL. Relationship between difficult tracheal intubation and obstructive sleep apnoea. Br J Anaesth. 1998 May;80(5):606-11. doi: 10.1093/bja/80.5.606. PMID 9691863
- [Result] Lee SJ, Lee JN, Kim TS, Park YC. The relationship between the predictors of obstructive sleep apnea and difficult intubation. Korean J Anesthesiol. 2011 Mar;60(3):173-8. doi: 10.4097/kjae.2011.60.3.173. Epub 2011 Mar 30. PMID 21490818
- [Result] Siyam MA, Benhamou D. Difficult endotracheal intubation in patients with sleep apnea syndrome. Anesth Analg. 2002 Oct;95(4):1098-102, table of contents. doi: 10.1097/00000539-200210000-00058. PMID 12351303